CLINICAL TRIAL: NCT01464671
Title: STATUS-PCI: Stable Angina Therapy With Angiomax® or Unfractionated Heparin for patientS Undergoing Percutaneous Coronary Intervention
Brief Title: Angiomax® or Unfractionated Heparin for Patients Undergoing Percutaneous Coronary Intervention
Acronym: STATUS PCI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: DSMB halted the study early due to futility. There were no safety concerns.
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Allen Jeremias, Associate Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 119778 (IRB ID)
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Stable Angina; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable | interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bivalirudin (Active Comparator): Anticoagulation during percutaneous coronary intervention
  Interventions: Drug: Bivalirudin; Drug: Heparin
- Unfractionated Heparin (Active Comparator): Anticoagulation during percutaneous coronary intervention
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Bivalirudin — Anticoagulation during percutaneous coronary intervention
  Other Names: Angiomax
  Arms: Bivalirudin
Drug: Heparin — Anticoagulation during percutaneous coronary intervention

SUMMARY:
The objective of the study is to assess the safety and efficacy of Angiomax® (bivalirudin) versus unfractionated heparin (UFH) in patients presenting with stable angina or silent ischemia (positive stress test without chest pain) that undergo percutaneous coronary intervention (PCI).

The primary endpoint of the study will be major and minor bleeding events, defined by the REPLACE-2 trial definition, during the index hospitalization and up to 30 days post discharge.

DETAILED DESCRIPTION:
The purpose of this study is to compare in a randomized, controlled, single-blinded, 1:1 fashion UFH versus bivalirudin in patients with stable angina pectoris or silent ischemia undergoing PCI.

Secondary study endpoints will include:

* Major adverse cardiac events (MACE) comprising of all cause mortality, myocardial infarction (MI), ischemia driven target vessel revascularization (TVR), and cerebral vascular accident (CVA).
* Net adverse clinical events (NACE) will be consistent of MACE plus major bleeding as defined by the REPLCE-2 criteria.
* Cardiac death in-hospital and up to 30 days post discharge.
* MI in-hospital and up to 30 days post discharge.
* CVA in-hospital and up to 30 days post discharge.
* Incidence of all-cause mortality at 6 months and 1 year.
* MACE at 6 months and 1 year.
* Incidence of acute (0-24 hours post procedure) stent thrombosis rates.
* Incidence of sub-acute (24 hours - 30 days) stent thrombosis rates.
* Length of hospital stay (LOS)
* Economic analysis (total cost during hospitalization) and up to 30 days post discharge.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is male or female ≥ 18 years of age.
2. The patient presents with stable angina pectoris, or silent ischemia (positive stress test without chest pain).
3. The patient is scheduled for coronary angiography, with possible angioplasty.
4. The patient is able to tolerate dual anti-platelet therapy with aspirin and clopidogrel for a minimum of 30 days and is on those medications at the time of the PCI (clopidogrel may be administered during PCI or within 30 minutes post PCI).
5. The patient is able and willing to conform to the requirements of the study and voluntarily signs an Informed Consent.
6. The patient does not present with any form of illness or condition that in the investigator's opinion would impair the results of the study.
7. Women of child bearing potential must have a negative urine or serum pregnancy test prior to enrollment.

Exclusion Criteria:

1. Patients in cardiogenic shock.
2. Patients with acute coronary syndrome, which includes unstable angina, non-ST-elevation MI or STEMI.
3. Known history of heparin-induced thrombocytopenia.
4. Contraindication to unfractionated heparin, bivalirudin, or any anticoagulant or antithrombotic pharmacological agent.
5. Any significant medical condition, which in the investigator's opinion, may interfere with the patient's optimal participation in the study.
6. Pregnant women or nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2009-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Bleeding events | 30 days
  The primary endpoint of the study will be major and minor bleeding events, defined by the REPLACE-2 trial definition during the index hospitalization and up to 30 days post discharge.

SECONDARY OUTCOMES:
MACE | 1 year
  Major adverse cardiac events (MACE) comprising of all cause mortality, myocardial infarction (MI), ischemia driven target vessel revascularization (TVR), and cerebral vascular accident (CVA).

CONTACTS AND LOCATIONS:
Overall Officials: Allen Jeremias, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States